CLINICAL TRIAL: NCT04328168
Title: Comparision Of The Effectiveness Of Conventional Physiotherapy After Botulinum Toxin Injection In Children With Cerebral Palsy
Brief Title: Comparision Of The Effectiveness Of Physiotherapy Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Ayşe Güç, Kayseri Education and Research State Hospital, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016/442
Record Dates: First submitted 2020-03-21; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Cerebral Palsy
Keywords: Botulinum-toxin, cerebral-palsy, robot-assisted therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: A total of 28 patients who were followed-up in our clinic and received botulinum toxin injection of lower extremities in the last month were randomized to two groups in the study. Group 1 received conventional physiotherapy and Group 2 received robot-assisted gait training.
Who Masked: Participant
Masking Description: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Active Comparator): Conventional Physiotherapy
  Interventions: Procedure: ROM exercises, stretching, positioning, gait training
- Group2 (Active Comparator): robot-assisted gait training
  Interventions: Procedure: by two physiotherapist under the supervision of a doctor

INTERVENTIONS:
Procedure: ROM exercises, stretching, positioning, gait training
  Arms: Group1
Procedure: by two physiotherapist under the supervision of a doctor
  Arms: Group2

SUMMARY:
A total of 28 patients who were followed-up in our clinic and received botulinum toxin injection of lower extremities in the last month were randomized to two groups in the study. Group 1 received conventional physiotherapy and Group 2 received robot-assisted gait training. The treatment period was 30 min/day, five sessions in a week, 15 sessions in total, for both groups. The study population was evaluated using range of joint motion evaluation chart, the Modified Ashworth Scale, The Gross Motor Function Classification System, The Berg Balance Scale, the functional independence measure for children, and the Edinburgh Visual Gait Score

DETAILED DESCRIPTION:
A total of 28 patients who were followed-up in our clinic and received botulinum toxin injection of lower extremities in the last month were randomized to two groups in the study. Group 1 received conventional physiotherapy and Group 2 received robot-assisted gait training. The treatment period was 30 min/day, five sessions in a week, 15 sessions in total, for both groups. The study population was evaluated using range of joint motion evaluation chart, the Modified Ashworth Scale, The Gross Motor Function Classification System, The Berg Balance Scale, the functional independence measure for children, and the Edinburgh Visual Gait Score.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4>, <16 with CP diagnosis
* Walking diffculties due to the spasticity of lower extremities,
* Level I-IV on the Gross Motor Function Classification System.

Exclusion Criteria:

* MAS Level IV spasticity, contractures, or rigidity in the lower extremities,
* A limb length inequality of >2 cm,
* Hypotonic CP,
* Having drug-related refractory epilepsy,
* Undergoing intrathecal baclofen pump surgery,
* Surgical interventions in the lower extremities in the last year,
* Scoliosis angle of >30°,
* Complicated osteoporosis (nontraumatic fracture...),
* Cardiovascular instability,
* GMFCS Level V,
* Metabolic disorder, genetic disease, neurodegenerative and neuromuscular diseases.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
The Gross Motor Function Classification System (GMFCS) | 3 weeks
  The Gross Motor Function Classification System or GMFCS is a 5 level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities.
The Edinburgh Visual Gait Scale (EVGS) | 3 weeks
  The Edinburgh visual gait score is an evaluative tool that uses software and video cameras to provide 3D video gait analysis as well as onscreen drawing and measurement tools to evaluate each portion of gait. The software will then generate a EVGS report, with illustrative images from the video if desired, in PDF format.

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) is not be available to other researchers.